CLINICAL TRIAL: NCT00121485
Title: The HeartMate II LVAS Pivotal Study Protocol, Destination Therapy
Brief Title: Thoratec HeartMate II Left Ventricular Assist System (LVAS) for Destination Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC010230-2
Record Dates: First submitted 2005-07-12; First posted 2005-07-21 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Congestive; Ventricular Dysfunction; Cardiomyopathies
Keywords: Heart-assist devices
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies | interventions — Heart-Assist Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HeartMate II (Experimental): Implantation of HeartMate II LVAS
  Interventions: Device: Left Ventricular Assist System (LVAS)
- HeartMate XVE (Active Comparator): Implantation of HeartMate XVE LVAS
  Interventions: Device: Left Ventricular Assist System (LVAS)

INTERVENTIONS:
Device: Left Ventricular Assist System (LVAS) — Implantation of left ventricular assist device for hemodynamic support
  Other Names: Thoratec; HeartMate II; ventricular assist

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Thoratec HeartMate II Left Ventricular Assist System (LVAS) as Destination Therapy in end-stage heart failure patients who do not qualify for cardiac transplantation.

The Destination Therapy indication for use was approved by FDA on January 20, 2010 (ref. PMA P060040/S005).

DETAILED DESCRIPTION:
The HeartMate II is a high speed, electric, axial flow, rotary blood pump. The pump drains blood from the left ventricular apex via a rigid inlet cannula and ejects into the aortic root via an outflow cannula joined to the aorta with an end to side anastomosis. Power and control of the pump are delivered through a percutaneous cable from the pump to the belt-worn System Driver.

The Destination Therapy trial is a prospective, randomized, unblinded, non-inferiority evaluation of the HeartMate II LVAS, compared to the HeartMate XVE.

ELIGIBILITY:
Inclusion Criteria:

The following are general criteria; more specific conditions are included in the study protocol:

* Subjects with advanced heart failure symptoms (NYHA Class IIIB or IV) who are:

  * On optimal medical management and are failing to respond; or
  * In Class III or Class IV heart failure and dependent on IABP and/or inotropes; or
  * Treated with ACE inhibitors or beta-blockers and found to be intolerant.
* Ineligible for cardiac transplant
* VO2max <=14 ml/kg/min
* LVEF <=25%

Exclusion Criteria:

The following are general criteria; more specific conditions are included in the study protocol:

* Evidence of, or risk factors for end-organ dysfunction that would make LVAS implantation futile
* Existence of factors that would adversely affect patient survival or function of the LVAS
* Intolerance to anticoagulant or antiplatelet therapies.
* Existence of any ongoing mechanical circulatory support other than intra-aortic balloon counterpulsation.
* Participation in any other clinical investigation that is likely to confound study results or affect study outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-02; Primary Completion 2009-06 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec Corporation
Locations (47):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Hospital @ University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Methodist Hospital, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts / New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital/Washington University, St Louis, Missouri
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Columbia Presbyterian Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Milton Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Hospital of University of PA, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Medical City Hospital Dallas, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - LDS Hospital (Intermountain Health Care), Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Medical School, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Hospital Royal Victoria / McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Result] Slaughter MS, Rogers JG, Milano CA, Russell SD, Conte JV, Feldman D, Sun B, Tatooles AJ, Delgado RM 3rd, Long JW, Wozniak TC, Ghumman W, Farrar DJ, Frazier OH; HeartMate II Investigators. Advanced heart failure treated with continuous-flow left ventricular assist device. N Engl J Med. 2009 Dec 3;361(23):2241-51. doi: 10.1056/NEJMoa0909938. Epub 2009 Nov 17. PMID 19920051
- [Result] Petrucci RJ, Rogers JG, Blue L, Gallagher C, Russell SD, Dordunoo D, Jaski BE, Chillcott S, Sun B, Yanssens TL, Tatooles A, Koundakjian L, Farrar DJ, Slaughter MS. Neurocognitive function in destination therapy patients receiving continuous-flow vs pulsatile-flow left ventricular assist device support. J Heart Lung Transplant. 2012 Jan;31(1):27-36. doi: 10.1016/j.healun.2011.10.012. PMID 22153550
- [Result] Park SJ, Milano CA, Tatooles AJ, Rogers JG, Adamson RM, Steidley DE, Ewald GA, Sundareswaran KS, Farrar DJ, Slaughter MS; HeartMate II Clinical Investigators. Outcomes in advanced heart failure patients with left ventricular assist devices for destination therapy. Circ Heart Fail. 2012 Mar 1;5(2):241-8. doi: 10.1161/CIRCHEARTFAILURE.111.963991. Epub 2012 Jan 26. PMID 22282104
- [Derived] Brisco MA, Sundareswaran KS, Milano CA, Feldman D, Testani JM, Ewald GA, Slaughter MS, Farrar DJ, Goldberg LR; HeartMate II Clinical Investigators. Incidence, risk, and consequences of atrial arrhythmias in patients with continuous-flow left ventricular assist devices. J Card Surg. 2014 Jul;29(4):572-80. doi: 10.1111/jocs.12336. Epub 2014 Apr 18. PMID 24750460

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HeartMate II | HeartMate XVE
Started | 134 | 66
Completed | 133 | 59
Not Completed | 1 | 7
Not completed — Not implanted | 1 | 5
Not completed — Crossover | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HeartMate II | HeartMate XVE | Total
Number analyzed (Participants) | 134 | 66 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12) | 63 (12) | 62.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 5 | 31
  Male | 108 | 61 | 169
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 0 | 2
  Hispanic | 4 | 0 | 4
  Black or African American | 24 | 16 | 40
  White | 101 | 48 | 149
  Other, unknown | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint
Description: Survival at two (2) years free of stroke, or reoperation to repair or replace the device
Time Frame: Patients' status at 2 years post-implant
Population: Primary Study Cohort (Intent to Treat)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 134 | 66
percentage of participants | 46 [38 to 55] | 11 [3 to 18]
Statistical Analysis 1: Comparison: HeartMate II vs HeartMate XVE; Primary endpoint is 2-yr survival free of stroke or re-operation to repair/replace the device. Patients are a success if composite endpoint achieved. Patients urgently transplanted due to device failure are failures. Patients electively transplanted after reversal of co-morbidity will be considered success if they achieve 2 years of survival from day of VAD implant and no stroke. HMII is a success if the proportion of HMII pts achieving the composite endpoint is equal to or better than HM XVE; Test type: Non-Inferiority or Equivalence — 200 patients (137 HMII and 67 XVE) provides 80% power (alpha= 0.05 (one-sided)) using a Blackwelder like analysis and a non-inferiority margin of 10%. The protocol specifies that once non-inferiority is proven, the data will be analyzed for superiority using closed testing methods; p = 0.00000025, Fisher Exact — Two (2) interim analysis were pre-specified in the protocol. The type I error rate was preserved at 5% by use of the O'Brien-Fleming spending function; Mean Difference (Final Values) = 35.7, 95% CI 2-sided [24.5 to 46.9]

2. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire(MLWHF)
Description: MLWHF is a validated instrument to self assess how heart failure and its treatment affect the key physical, emotional, social and psychological dimensions of quality of life. The instrument is made up of 21 items that assess the patient's perception of these dimensions on a scale ranging from no (0) to very much (5). The total MLWHF score is calculated by adding the scores for all 21 items (range, 0-105). A lower score indicates a better quality of life. The patients' scores at Baseline, 1, 3, 6 and 12 Months post-implant are presented and indicate improved quality of life.
Time Frame: Baseline, Months 1,3,6,12
Population: Primary Study Cohort (As Treated)
Measure: Mean (Standard Deviation); unit: Units on a MLWHF Score scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 133 | 59
Units on a MLWHF Score scale
  Baseline | 75.2 (17.7) | 76.3 (18.1)
  1 Month | 62.8 (23.7) | 59.1 (26.5)
  3 Months | 37.4 (22.2) | 43.6 (23.8)
  6 Months | 36.5 (23.3) | 46.4 (21.0)
  12 Months | 33.6 (22.1) | 41.2 (21.4)

3. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: KCCQ is a validated instrument to self assess quality of life including physical function and social function. Scores are calculated based on responses to the questionnaire, on a scale from 0-100. The higher the score, the better the quality of life. The patients' scores at Baseline, 1, 3, 6 and 12 Months are presented and indicate improved quality of life.
Time Frame: Baseline, Months 1, 3, 6, 12
Population: Primary Study Cohort (As Treated)
Measure: Mean (Standard Deviation); unit: Units on a KCCQ score scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 133 | 59
Units on a KCCQ score scale
  Baseline | 27.4 (16.3) | 26.5 (17.4)
  1 Month | 41.8 (20.3) | 38.9 (23.2)
  3 Months | 63.4 (18.5) | 56.7 (21.1)
  6 Months | 64.2 (20.4) | 55.5 (21.5)
  12 Months | 65.9 (20.0) | 61.1 (20.4)

4. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: NYHA relates symptoms to every day activities and patients quality of life. Class 1 = no limitations on physical activity Class 2 - slight limitation of physical activity Class 3 - marked limitation of physical activity Class 4 = unable to carry out any physical activity without discomfort
Time Frame: Baseline, Months 1, 6, 12
Population: Primary Study Cohort (As Treated)
Measure: Number; unit: percentage of participants in each class
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 133 | 59
percentage of participants in each class
  Baseline NYHA Class I - II | 0 | 0
  Baseline NYHA Class III - IV | 100 | 100
  1 Month NYHA Class I - II | 45 | 45
  1 Month NYHA Class III - IV | 56 | 55
  6 months NYHA Class I - II | 79 | 73
  6 Months NYHA Class III - IV | 19 | 27
  12 Months NYHA Class I - II | 76 | 61
  12 Months NYHA Class III - IV | 24 | 39

5. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The Six Minute Walk Test(6MWT) measures the distance that a patient can walk in a period of 6 minutes. The distance walked is measured in meters. This test measures the patients' functional status. The more meters a patient can walk over baseline indicates improvement in functional status.
Time Frame: Baseline, Months 1, 3, 6, 12
Population: Primary Study Cohort (As Treated)
Measure: Mean (Standard Deviation); unit: Distance (meters)
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 133 | 59
Distance (meters)
  Baseline | 182.5 (140.6) | 172.2 (107.7)
  1 Month | 244.2 (179.2) | 236.0 (134.1)
  3 Months | 316.5 (191) | 291.0 (136.5)
  6 Months | 377.2 (252.7) | 339.7 (134.4)
  12 Months | 317.6 (163.6) | 307.6 (144.9)

6. Secondary Outcome: Functional Status (Patient Activity Score)
Description: Metabolic Equivalent Score (METs). Ranges: Very Low, Low, Moderate, High, Very High
Time Frame: Baseline, Months 1, 3, 6, 12
Population: Primary Study Cohort (As Treated)
Measure: Number; unit: percentage of participants
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 133 | 59
percentage of participants
  Baseline (Very Low, Low) | 95 | 94
  Baseline (Moderate, High, Very High) | 5 | 6
  1 Month (Very Low, Low) | 86 | 90
  1 Month (Moderate, High, Very High) | 14 | 10
  3 Months (Very Low, Low) | 53 | 58
  3 Months (Moderate, High, Very High) | 47 | 42
  6 Months (Very Low, Low) | 45 | 56
  6 Months (Moderate, High, Very High) | 55 | 44
  12 Months (Very Low, Low) | 39 | 62
  12 Months (Moderate, High, Very High) | 61 | 38

7. Secondary Outcome: Reoperations
Description: The number of additional surgeries after the initial pump implant. Data is presented as the percentage of patients who required a reoperation for pump replacement or repair, bleeding or other reasons
Time Frame: Patients were followed until outcome or up to 2 years post-implant, whichever came first
Measure: Number; unit: percentage of participants
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 133 | 59
percentage of participants
  Pump Replacement | 9 | 32
  Pump Repair | 0 | 1.7
  Bleeding | 44.4 | 23.7
  Other | 60.2 | 54.2

8. Secondary Outcome: Neurocognitive Assessments, Clock Drawing
Description: Clock drawing is a measure of visual-spatial integrity, visual motor skills and organizational ability. The drawing was administered with the command version with no time restraint. The clock is scored from 1-10, with 10 a better score.
Time Frame: Baseline (1 month), 6 months
Population: Patients enrolled at 12 representative study sites participated in the neurocognitive testing. These study sites were selected based on their historic implant rates to represent high, medium and low enrolling centers.
Measure: Median (Full Range); unit: units on a scale
Groups:
- HeartMate XVE: Implantation of HeartMate XVE
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 44 | 16
units on a scale
  Clock drawing, baseline | 9.0 [4 to 10] | 8.5 [4 to 10]
  Clock drawing, 6 months | 9 [4 to 10] | 9 [4 to 10]

9. Secondary Outcome: Neurocognitive Assessments, Wechsler Memory Scale-III (WMS-LM and WMS-LM Delayed)
Description: The WMS-LM is a measure of auditory attention and memory. This contextual memory task requires patients to recall a passage read by the examiner. Their memory tasks are avoided during the intervening time so as not to disrupt recall. The WMS-LM test provides a comparision for immediate recall and the WMS-LM Delayed provides a comparison for recall that is delayed 30 minutes. The test is scored in a range from 0-50, where the higher score is considered better
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 46 | 16
units on a scale
  WMS-LM, Baseline | 19.5 [4 to 32] | 20.0 [3 to 33]
  WMS-LM, 6 months | 24.0 [5 to 45] | 14.0 [5 to 29]
  WMS-LM Delayed, Baseline | 16 [4 to 28] | 12.5 [1 to 31]
  WMS-LM Delayed, 6 months | 18.5 [1 to 36] | 13 [1 to 27]

10. Secondary Outcome: Neurocognitive Assessments, Wechsler Memory Scale-III Visual Reproduction (WMS-VR and WMS-VR Delayed)
Description: The WMS-VR is a measure of visual memory. This is a graphic memory task requiring both immediate recall and after a 30 minute delay (WMS-VR Delayed). The scoring range is 0-104 where the higher score is better.
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 44 | 16
units on a scale
  WMS-VR, Baseline | 71.1 [13 to 102] | 76.0 [21 to 101]
  WMS-VR, 6 months | 79 [27 to 104] | 68 [5 to 100]
  WMS-VR Delayed, Baseline | 32 [2 to 90] | 37 [6 to 98]
  WMS-VR Delayed, 6 months | 50.5 [8 to 93] | 38.0 [4 to 97]

11. Secondary Outcome: Neurocognitive Assessments, Wechsler Adult Intelligence Test-III, Block Design (WAIS Block)
Description: The WAIS block is a measure of visual spatial and visual motor ability. The patient is given a stimulus configuration to replicate with red and white blocks while being timed, first starting with four blocks and progressing to a nine block configuration. Performance is scored on time upon full completion of the task with a maximum of 68 points. The higher the score, the better.
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 43 | 16
units on a scale
  WAIS Block, Baseline | 29.0 [12 to 50] | 25.5 [5 to 50]
  WAIS Block, 6 months | 31.0 [10 to 64] | 28.0 [12 to 44]

12. Secondary Outcome: Neurocognitive Assessments, Boston Naming Test
Description: Fifteen pictures of objects are presented to the patient. The patient is asked to name the object without prompting. A Correct identification represents one point. This test is designed to test language. Scores are from 0-15, higher being better.
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 45 | 16
units on a scale
  Boston Naming, Baseline | 14.0 [4 to 15] | 14.0 [9 to 15]
  Boston Naming, 6 months | 14.0 [6 to 15] | 13 [10 to 15]

13. Secondary Outcome: Wechsler Adult Intelligence Test-III, Digit Symbol (WAIS Digit)
Description: The WAIS Digit is a measure of visual motor speed and abstracting ability. The patient is given the numbers one to nine with an associated symbol. Performance is scored on time with correct amount completed with a maximum of 133 points, where higher is better.
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 43 | 15
units on a scale
  WAIS Digit, Baseline | 45 [9 to 89] | 31 [4 to 85]
  WAIS Digit, 6 months | 45 [13 to 84] | 34 [10 to 73]

14. Secondary Outcome: Neurocognitive Assessments, Trail Making A
Description: This is a visual motor task measuring processing speed. The patient is required to draw a line between sequential numbers while being timed to completion. The score is time to completion in seconds and lower score is better.
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: Units measured in seconds
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 42 | 14
Units measured in seconds
  Trail Making A, Baseline | 45.5 [23 to 148] | 52.0 [19 to 119]
  Trail Making A, 6 months | 44.0 [16 to 77] | 52 [25 to 130]

15. Secondary Outcome: Neurocognitive Assessments, Trail Making B
Description: This is a visual motor task measuring processing speed and executive functions. The patient is required to draw a line between alternating sequential numbers and letters while being timed to completion. Testing scores are time to completion in seconds with lower score being better.
Time Frame: Baseline (1 month), 6 months
Population: as for outcome 8
Measure: Median (Full Range); unit: Units measured in seconds
Arm/Group | HeartMate II | HeartMate XVE
Number analyzed (Participants) | 41 | 14
Units measured in seconds
  Trail Making B, Baseline | 122.0 [30 to 495] | 152.5 [43 to 403]
  Trail Making B, 6 months | 117.0 [33 to 423] | 188.5 [55 to 420]

ADVERSE EVENTS:
Time Frame: Patients were followed until outcome (transplanted, explanted, expired, withdrawn), for an average of 1.2 years
Description: All serious adverse events for duration of study are listed below
Arm/Group | HeartMate II | HeartMate XVE
Serious Adverse Events (participants affected / at risk) | 129/133 | 58/59
Other Adverse Events (participants affected / at risk) | 86/133 | 42/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartMate II (N=133) | HeartMate XVE (N=59)
Bleeding (All serious events) (Blood and lymphatic system disorders) | 102 (278) | 41 (70) — events that cause death, reoperations, permanent injury or necessitate transfusion of >2 units of PRBC within 24 hours
Bleeding requiring surgery (Surgical and medical procedures) | 40 (50) | 9 (12)
Stroke (Nervous system disorders) | 24 (27) | 8 (9) — neurological deficit lasting more than 24 hours or lasting 24 hours or less with a brain imaging study showing new infarction
Other neurological (Nervous system disorders) | 27 (32) | 9 (11) — any new, temporary or permanent, focal or global neurological deficit including TIA, metabolic encephalopathy, seizure, etc
Local Infection (Infections and infestations) | 40 (60) | 19 (30) — Localized non-device related infections
Drive Line Infection (Infections and infestations) | 39 (75) | 14 (22) — infection of the drive line
Pocket Infection (Infections and infestations) | 12 (19) | 8 (10) — Infection of the pump pocket
Pump Housing (Infections and infestations) | 1 (1) | 2 (2) — Infection of the pump housing
Sepsis (Infections and infestations) | 48 (80) | 26 (45) — a systemic response to a serious infection, usually manifested by fever, tachycardia, tachypnea, leukocytosis and vasodilatation requiring use of IV antimicrobial therapy
Right Heart Failure (Inotropes) (Cardiac disorders) | 27 (29) | 16 (19) — Need for inotropic support for > 14 days after implant
Right Heart Failure (RVAD) (Cardiac disorders) | 5 (5) | 3 (3) — the need for RVAD
Peripheral Thromboembolism (Vascular disorders) | 14 (21) | 6 (6) — Any thrombus or thrombo-embolism in the pulmonary or systemic circulations confirmed by standard clinical and laboratory testing, or operative findings, or autopsy findings, or that requires empirical intervention
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 47 (61) | 24 (33) — Impairment of respiratory function requiring reintubation and/or tracheostomy at any time or the inability to discontinue ventilatory support after 6 days of VAD support
Cardiac Arrhythmia (Cardiac disorders) | 62 (110) | 21 (30) — any arrhythmia that requires intervention
Renal Failure (Renal and urinary disorders) | 21 (21) | 14 (14) — require renal replacement therapy (CVVHD or dialysis) that was not required prior to implant
Hepatic Dysfunction (Hepatobiliary disorders) | 3 (3) | 0 (0) — liver function studies that are greater than three times the baseline values in any two of the three liver function studies (total bilirubin, AST and ALT)
Device Thrombosis (Blood and lymphatic system disorders) | 5 (5) | 0 (0) — thrombus in device or conduits with symptoms of impaired pump performance (e.g. decreased pump flow, need increase speed, increased power, hemolysis) or need for thrombolytic or surgical intervention
Hemolysis (Blood and lymphatic system disorders) | 5 (5) | 0 (0) — two consecutive PHgb values above 40 mg/dl and a LDH value above 1,000mg/dl during the same time
Psychological (Psychiatric disorders) | 4 (4) | 0 (0) — disturbance in thinking, emotion or behavior that causes substantial impairment in functioning or marked subjective distress requiring intervention
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Confirmed Malfunctions (Cardiac disorders) | 30 (39) | 12 (14)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartMate II (N=133) | HeartMate XVE (N=59)
Bleeding (Blood and lymphatic system disorders) | 16 (121) | 10 (43)
Local Infection (Infections and infestations) | 25 (100) | 8 (25)
Cardiac Arrhythmia (Cardiac disorders) | 13 (35) | 14 (24)
Psychological (Psychiatric disorders) | 4 (7) | 4 (4)
Confirmed Malfunctions (Cardiac disorders) | 28 (73) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No